CLINICAL TRIAL: NCT06725199
Title: Metabolomic Profiling Based on Nuclear Magnetic Resonance in Fibromyalgia Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: hatice kübra aşık (Other)
Collaborators: University of Beykent (Other); Bezmialem Vakif University (Other)
Responsible Party: Sponsor-Investigator, hatice kübra aşık, assistant professor, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: E-80929729-000-212940150
Record Dates: First submitted 2024-12-04; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Patients with Clinical Complaints of Fibromyalgia Among the Patients Applying to the Outpatient Clinic; Fibromyalgia Syndrome
Keywords: fibromyalgia; metabolomics profiling
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy group: Blood and urine samples taken from completely healthy individuals will be examined.
- Fibromyalgia group: Blood and urine samples taken from individuals diagnosed with fibromyalgia will be examined

SUMMARY:
Evaluation of sera of fibromyalgia patients in terms of energy metabolism function and possible alterations in metabolism predisposing to various degenerative/proliferative diseases.

DETAILED DESCRIPTION:
1. Full name of the study: Nuclear Magnetic Resonance Based Metabolomic Profiling in Fibromyalgia Patients
2. Aim and importance of the study (primary aim, secondary aims, if any):

   Determination and quantitation of metabolites and enzyme activities by NMR in fibromyalgia patients, changes in citrate, isocitrate, alpha ketoglutarate, alpha ketoglutarate, succinyl CoA, fumarate, malate, glutamate, G-6 PD, phosphogluconate, glyceraldehyde 3 P and oxaloacetate values, especially in energy metabolism in these patients and evaluation of their clinical usefulness will be investigated.
3. Expected benefits and risks of the research:

   Fibromyalgia is defined as a chronic syndrome of unknown cause characterized by widespread body pain, fatigue, sleep disturbance, impaired cognitive functioning and anxiety, and possible causes include genetic, neurological, psychological, sleep-related and immunological factors. The disease is 6-9 times more common in women. The diagnosis of fibromyalgia, which has been defined as a true syndrome since the publication of the 1990 classification criteria of the American College of Rheumatology (ACR), is difficult due to the subjectivity of the symptoms, the fact that the evaluation is based on patient reports and the lack of objective diagnostic tests to confirm the diagnosis. The diagnostic criteria for fibromyalgia, which was first described in the 19th century and is the most common rheumatic disease after osteoarthritis, are in constant change. In addition to the difficulty in the diagnosis of the disease, the physiopathology is not fully understood and a specific target for treatment has not been determined.

   The number of metabolomic studies in serum and urine analyses of patients with fibromyalgia is limited and in order to fill this gap, we will use Bruker 500 MHertz NMR device with an experienced team to examine metabolite determination and quantitation, enzyme activities and especially energy metabolism in Fibromyalgia patients. Thus, it will be investigated whether there is a predisposition to degenerative or proliferative diseases due to acceleration or decrease in energy metabolism in Fibromyalgia patients. According to our literature review, there are no studies investigating both enzymes and metabolites together in fibromyalgia patients.

   In the published work of researchers, NMR is often used for structure analysis. Quantitative NMR (qNMR), on the other hand, is under development to expand the range of metabolites it can detect in body fluids (to capture low concentrations of substances). qNMR started with very old studies and sub-techniques are being optimized to provide high sensitivity. With the developing technology, this spectrum will expand and in the future, hundreds of metabolites can be determined using a single reference. Although NMR equipment is available in a limited number of universities in our country, we have determined that there is no group working for quantitative analysis as a result of our research. We aim to put our theoretical knowledge into practice with the experience and knowledge of the faculty members of Bezmi Alem Vakıf University Faculty of Medicine within our project.

   As a starting point for our qNMR studies, we chose fibromyalgia disease, where the number of daily samples reaching our hospital is quite high. In addition, we found that clinical studies on the subject are quite limited. In this sense, the investigators is unique in that it will provide a holistic metabolic profiling in fibromyalgia patients and provide data on adults.

   The most important problem with the NMR technique is the high costs during the installation of the device, then with low operating costs, the desired analyzes can be performed easily and at low cost in the presence of reference materials and software required for data analysis. We aim to perform quantification of metabolites in body fluids on the NMR device, which has already been installed and is currently in operation at Bezmi Alem Vakıf University. As a starting point, we chose fibromyalgia disease, for which quantitative NMR analysis is very rare in the literature. In terms of sample preparation/analysis procedure for quantitative NMR analyses, it is planned to study serum and urine, which are the first standardized body fluid samples, and samples belonging to the patient population and healthy volunteers. According to the peaks obtained in the NMR spectrum, metabolite identification will be made and quantitation of these metabolites will be performed with the software to be provided for the study.
4. Type, scope and design of the planned study:

   In this prospective two-group study, metabolite identification will be performed according to the peaks obtained in the NMR spectrum in 50 patients with clinically diagnosed fibromyalgia and 50 healthy volunteers and it is aimed to perform the quantitation of these metabolites with the software to be provided for the study.
5. Number of patients and volunteers to be included in the study, their qualifications and rationale for selection:

   The investigators will be conducted between January 1, 2024 and December 1, 2024 with 50 patients with a diagnosis of fibromyalgia between the ages of 18-65 who meet the inclusion and exclusion criteria of the investigatorsand 50 healthy volunteers. The prior power analysis of the study was performed using the "G. Power-3.1.9.2" program. Means in calculations: Wilcoxon singed-rank test (one sample case) effect size 0.50, alpha 0.05, power 0.90, number of groups 1, number of measures:2, total sample was calculated as 38. A total of 38 patients were planned to be included in the study
6. Parameters to be analyzed:

   Measurement of citrate, isocitrate, alpha ketoglutarate, succinyl CoA, fumarate, malate, glutamate, G-6 PD, phosphogluconate, glyceraldehyde 3 P and oxaloacetate levels by NMR technique
7. Where and by whom the parameters will be checked: The study will be conducted by Specialist Dr. Hatice Kübra Aşık in the outpatient clinic of the Physical Medicine and Rehabilitation Clinic of Private Beykent Hospital. Dr. Hatice Kübra Aşık and biochemical tests will be performed by Prof. Dr. Yıldız Atamer at the Biochemistry Department of Private Beykent Hospital.
8. Which of the parameters to be used in the study are routine for that disease group and which are specific to the study:

   Measurement of citrate, isocitrate, alpha ketoglutarate, succinyl CoA, fumarate, malate, glutamate, G-6 PD, phosphogluconate, glyceraldehyde 3 P and oxaloacetate levels by NMR technique not routine for this disease but will be studied in this group for scientific research purposes
9. Projected duration of work, start and end dates: March 1, 2024 - December 1, 2024
10. Inclusion, exclusion and withdrawal criteria:

    Inclusion criteria:

    Female patients aged 18-65 years Patients with clinical complaints of fibromyalgia (widespread pain, weakness, fatigue, sleep problems, anxiety, restriction of movement, etc.) among the patients applying to the outpatient clinic

    Exclusion criteria:

    Viral or bacterial infections, Systemic diseases (diabetes mellitus, hypertension, chronic renal failure, hypo-hyperthyroidism) Patients taking antidepressants or medication, Patients with abnormal laboratory results (erythrocyte sedimentation rate, biochemical or serologic parameters, and thyroid function tests), Smokers and alcohol users, Patients with rheumatic arthritis and systemic lupus erythematosus were excluded.

    Those who received treatment for tumor
11. Study termination criteria: The study is planned to be terminated after the completion of the 50 patients and 50 healthy volunteers required for the study.
12. In the evaluation of the data to be obtained as a result of the research statistical methods to be used:

IBM SPSS (Statistical Package for the Social Sciences) Statistics for Windows, Version 25.0. Armonk, NY: IBM Corp. will be used. In the descriptive statistics of the data, mean and standard deviation values will be used in parametric tests; median values, minimum and maximum values will be used in nonparametric tests.

The distribution of variables will be checked by Kolmogorov-Smirnov test. Paired t test will be used for repeated measurements with normal distribution, while Wilcoxon test will be used for non-normally distributed data. Results will be evaluated at 95% confidence interval and p<0.05 is defined as statistical significance.

1. Malatji BG, Meyer H, Mason S, et al. NMR metabolomics studies of selected patients and controls based on a diagnostic biomarker profile for fibromyalgia syndrome. BMC Neurology (2017), 17:88
2. Hsu W-H, Lee C-H, Chao Y-M, et al. ASIC3-dependent metabolomic profiling of serum and urine in fibromyalgia mouse model Scientific Reports, (2019), 9:12123.
3. Clos-Garcia M, Andrés-Marin N, Fernández-Eulate G, et al. Gut microbiome and serum metabolome analyses identify molecular biomarkers and altered glutamate metabolism in fibromyalgia. EBioMedicine (2019), 46:499-511.
4. Hackshaw KV, Aykas DP, Sigurdson GT, et al. Metabolic fingerprinting for the diagnosis of fibromyalgia and other rheumatologic disorders. J. Biol. Chem. (2019), 294(7):2555-2568.
5. Hsu W-H, Han D-S, Ku W-C, et.al. Metabolomic and proteomic characterization of sng and pain phenotypes in fibromyalgia. Eur J Pain, (2022), 26:445-462.
6. Victoria Menzies, Angela Starkweather, Yingwei Yao, et al. Metabolomic Differences in Women With and Without Fibromyalgia. Clin Transl Sci (2020) 13, 67-77.
7. Bal SH, Budak F. Overview of Genomics, Proteomics Concepts and Application Areal Journal of Uludag University Faculty of Medicine, 39 (1)65-69, 2013.
8. Başaran E, Aras S, Cansaran-Duman D. General Outlook and Applications of Genomics, Proteomics and Metabolomics.Turkish Journal of Hygiene and Experimental Biology 2010; 67 (2): 85-96.
9. Dogan HO. Untargeted Metabolomics Analysis. Sivas Biochemistry Days, November 2-5, 2016.
10. Marques AP, Santo ASE, Berssaneti AA, Matsutani LA, Yuan SLK. Prevalence of fibromyalgia: literature review update. Rev Bras Reumatol. 2017;57(4):356-363.
11. Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Häuser W, Flub E, et al. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017;76(2):318-328.

ELIGIBILITY:
Inclusion Criteria:

patients aged 18-65 years Patients with clinical complaints of fibromyalgia

Exclusion Criteria:

Viral or bacterial infections, Diabetes mellitus, Hypertension, Chronic renal failure, Hypo-hyperthyroidism) Patients taking antidepressants or medication, Smokers and alcohol users, Patients with rheumatic arthritis and systemic lupus erythematosus were excluded.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: patients aged 18-65 years Patients with clinical complaints of fibromyalgia and control group (healthy)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Metabolomic Profiling | September 2024- February 2025
  Biochemical enzymes will be measured by NMR techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Beykent, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
In this prospective two-group study, metabolite identification will be performed according to the peaks obtained in the NMR spectrum in 50 patients with clinically diagnosed fibromyalgia and 50 healthy volunteers and it is aimed to perform the quantitation of these metabolites with the software to be provided for the study.
  Measurement of citrate, isocitrate, alpha ketoglutarate, succinyl CoA, fumarate, malate, glutamate, G-6 PD, phosphogluconate, glyceraldehyde 3 P and oxaloacetate levels by NMR technique.
  Measurement of citrate, isocitrate, alpha ketoglutarate, succinyl CoA, fumarate, malate, glutamate, G-6 PD, phosphogluconate, glyceraldehyde 3 P and oxaloacetate levels by NMR technique not routine for this disease but will be studied in this group for scientific research purposes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Malatji BG, Meyer H, Mason S, Engelke UFH, Wevers RA, van Reenen M, Reinecke CJ. A diagnostic biomarker profile for fibromyalgia syndrome based on an NMR metabolomics study of selected patients and controls. BMC Neurol. 2017 May 11;17(1):88. doi: 10.1186/s12883-017-0863-9. PMID 28490352